CLINICAL TRIAL: NCT01302223
Title: Keratinocyte Growth Factor, Interleukin 1 Beta, 6, 8, 10, 12 and Tumor Necrosis Factor Alpha in Burned Patients.
Brief Title: Keratinocyte Growth Factor and Cytokines in Burns.
Status: Completed | Type: Observational
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, ALFREDO GRAGNANI FILHO, Associated Professor, Federal University of São Paulo
Other Study IDs: KGF and Cytokines in Burns
Record Dates: First submitted 2011-02-23; First posted 2011-02-24 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Burns; Growth Factors, Combined Defect of; Inflammation; Cytokine Storm
Keywords: burns; Growth Factors, Combined Defect of; inflammation; Cytokine Storm
MeSH Terms: conditions — Burns; Growth Factors, Combined Defect of; Inflammation; Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Normal skin will be collected at first burned patient debridment and send to Cell Culture Laboratory to start fibroblast and queratinocyte culture.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Minor Burns: Total burn surface area less than 5% of second and third degree.
- Major Burns.: Total Burn Surface Area more than 25% of second and third degree, and less than 50%.

SUMMARY:
KERATINOCYTE GROWTH FACTOR AND CYTOKINES IN SKIN BURNS.

INTRODUCTION: Intense inflammatory responses are activated by burns that affect a large total body surface area. Changes in plasma levels of cytokines after burns occur before metabolic abnormalities unsettle the patient. So it may be possible to develop therapeutic interventions that may attenuate the acute inflammatory response by decreasing the expression of these cytokines. The importance of growth factors in the healing process was demonstrated in cultured keratinocytes and fibroblasts. The keratinocyte growth factor (KGF) is a growth factor active in the repair of wounds, being the most potent stimulator of mitotic cells.

PURPOSE: To assess the level of keratinocyte growth factor (KGF) and IL-1ß, IL-6, IL-8, IL-10, IL-12 and TNF-alfa of patients with burns produced by cultured primary dermal fibroblasts and the gene expression.

METHODS: 10 patients will be include (05 patients in the study group and 05 patients in the control group) admitted to the Burns Care Unit of the Discipline of Plastic Surgery, Federal University of São Paulo (UNIFESP) between 25% and 50% of total body surface area (TBSA), deep second-degree or third degree, with need to perform surgical debridement. The control group will be constituted by patients with less than 5% of TBSA, deep second-degree or third degree, with need to perform surgical debridement. The authors will evaluate the levels of IL-1ß, IL-6, IL-8, IL-10, IL-12p70 and tumor necrosis factor alpha (TNF-alfa) in samples of the culture media of primary dermal fibroblasts of patients selected using flow cytometry. The level of keratinocyte growth factor (KGF), in the same samples will be evaluated by ELISA. The keratinocyte growth factor (KGF) and TNF-alfa gene expression will be evaluated in the culture of primary dermal fibroblasts from the same patients. The gene expression of KGF and cytokines will be done by qRT-PCR and RT-PCR array. The experiments will be done in duplicate.

DETAILED DESCRIPTION:
KERATINOCYTE GROWTH FACTOR AND CYTOKINES IN SKIN BURNS.

INTRODUCTION: Intense inflammatory responses are activated by burns that affect a large total body surface area. Changes in plasma levels of cytokines after burns occur before metabolic abnormalities unsettle the patient. So it may be possible to develop therapeutic interventions that may attenuate the acute inflammatory response by decreasing the expression of these cytokines. The importance of growth factors in the healing process was demonstrated in cultured keratinocytes and fibroblasts. The keratinocyte growth factor (KGF) is a growth factor active in the repair of wounds, being the most potent stimulator of mitotic cells.

PURPOSE: To assess the level of keratinocyte growth factor (KGF) and IL-1ß, IL-6, IL-8, IL-10, IL-12 and TNF-alfa of patients with burns produced by cultured primary dermal fibroblasts and the gene expression.

METHODS: 10 patients will be include (05 patients in the study group and 05 patients in the control group) admitted to the Burns Care Unit of the Discipline of Plastic Surgery, Federal University of São Paulo (UNIFESP) between 25% and 50% of total body surface area (TBSA), deep second-degree or third degree, with need to perform surgical debridement. The control group will be constituted by patients with less than 5% of TBSA, deep second-degree or third degree, with need to perform surgical debridement. The authors will evaluate the levels of IL-1ß, IL-6, IL-8, IL-10, IL-12p70 and tumor necrosis factor alpha (TNF-alfa) in samples of the culture media of primary dermal fibroblasts of patients selected using flow cytometry. The level of keratinocyte growth factor (KGF), in the same samples will be evaluated by ELISA. The keratinocyte growth factor (KGF) and TNF-alfa gene expression will be evaluated in the culture of primary dermal fibroblasts from the same patients. The gene expression of KGF and cytokines will be done by qRT-PCR and RT-PCR array. The experiments will be done in duplicate.

Key words: burns, cytokines, inflammation, keratinocyte growth factor, fibroblasts.

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* More than 18 years of age
* Burned patient
* Burned debridement necessary
* Inpatient of Burn Center of Federal University of São Paulo
* More than 25% and less than 50% of TBSA (group major burns)
* Less than 5% of TBSA (group minor burns)

Exclusion Criteria:

* Not interest in participating in research
* Not acceptance of surgical procedure
* Previous Skin disease
* Clinical disease that directly interferes with wound healing

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: ACUTE BURNED PATIENTS
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Keratinocyte Growth Factor | cultured cells at second passage
  Level of KGF in cultured fibroblasts at second passage in media culture and qRT-PCR and RT-PCR array.

SECONDARY OUTCOMES:
Interleucin 1 beta, 6, 8, 10, 12 and tumor necrosis factor alfa | cultured fibroblasts at second passage
  Level of cytokines in cultured fibroblasts at second passage in media culture and qRT-PCR and RT-PCR array.

CONTACTS AND LOCATIONS:
Overall Officials: ALFREDO GRAGNANI FILHO, MD, PhD, Principal Investigator — UFSaoPaulo; LYDIA M FERREIRA, MD Full Prof, Study Chair — UFSaoPaulo
Locations (1):
- Burn Center of Federal University of Sao Paulo, São Paulo, São Paulo, Brazil